CLINICAL TRIAL: NCT03665649
Title: Biomedical Study of Toxicity, Biodistribution, Expression and Cellular Characterization of Autologous CD133+ Stem Cells From Donors of Hematopoietic Progenitors (IGX1) in Murine Model With Asherman-induced Syndrome.
Brief Title: Pre-clinical Endometrial Tissular Renovation Study
Acronym: PreENTIRE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Igenomix (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IGX1-ASM-XS-18-06
Record Dates: First submitted 2018-09-07; First posted 2018-09-11 (Actual); Last update posted 2019-07-17 (Actual); Status verified 2019-07

CONDITIONS: Asherman Syndrome
Keywords: Asherman Syndrome; Bone marrow-derived stem cells; Endometrial regeneration; Assisted reproduction techniques; Endometrial physiopathology; CD133+; Endometrial atrophy; Endometrial thickness
MeSH Terms: conditions — Gynatresia; Macular Dystrophy, Retinal, 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CD133+ human donors (Other): CD133+ cells isolation
  Interventions: Procedure: CD133+ cells isolation

INTERVENTIONS:
Procedure: CD133+ cells isolation — Hematopoietic precursors from human donors will be mobilized by administering Colony Stimulating Factors (G-CSF) for 5 days (according to the clinical standard administration) and subsequently CD133+ cells will be isolated and transferred in a murine model.

SUMMARY:
The endometrium is a tissue with high capacity of renewal ("self-renewal"). This process is regulated by stem cells. Recent studies have shown that bone marrow-derived stem cells (BMDSCs) contribute to tissues and organs regeneration, including the murine and human endometrium. Additionally, BMDSCs have the ability to differentiate into functional endometrial and stromal epithelial cells.

Asherman's Syndrome (AS) also referred to as intrauterine adhesions (AIU), is an acquired uterine condition characterized by the formation of adhesions inside the uterus. In many cases the front and back walls of the uterus stick to one another. Most patients with AS have menstrual abnormalities, pelvic pain, recurrent miscarriage, and infertility, and psychological disorders. Currently, hysteroscopy is considered the gold standard of methods for the diagnosis of intrauterine adhesions. However, it has a limited capacity for treatment, especially in moderate or severe cases in which permanent infertility can occur. For the first time, our investigation group demonstrated the possibility of regenerating endometrial tissue through bone marrow-derived stem cells (Santamaria et al., 2016).

This project aims to determine the safety, tolerability and biodistribution of IGX1 (CD133+ cells selected after mobilization and collection of peripheral blood progenitor cells - CPSP) afte rthe intraarterial injection in rats with induced Asherman's Syndrome.

Therefore, the focus of this project is to satisfy the preclinical requirements set out by the the AEMPS (Agencia Española de Medicamentos y Productos Sanitarios) in relation to the Phase I/II clinical trial "Phase I-II clinical trial of advanced, prospective, open, non-randomized, uncontrolled (before-after study), explanatory, multicentre cell therapy , national, intervention with a single treatment group in patients of reproductive age with gestational desire diagnosed with Asherman's Syndrome grade II, III or IV, treated by autologous non-expanded bone marrow stem/progenitor cells selected (IGX1)" (IGX1-ENT-XS-16-01)

DETAILED DESCRIPTION:
The endometrium is the tissue that lines the inside of the uterine cavity and whose function is to enable implantation of the embryo at the right moment. When implantation of the embryo does not occur, the endometrium is partially destroyed and menstruation takes place, producing a new generation of tissue in the next menstrual cycle. It is therefore a high dynamic tissue undergoing changes of growth, differentiation and shedding every 28 days during 400-500 cycles during a woman's reproductive lifetime. This level of tissue regeneration is comparable to other tissues with high cellular turnover, such as epidermis, gut epithelium and bone marrow. This highly regenerative self-renewal capacity of the endometrium seems to be regulated by stem cells. An increased number of studies about endometrium-derived stem cells have been published in the last years. Furthermore, bone marrow-derived stem cells (BMDSCs) have been shown to contribute to the repair and regeneration of tissues and organs, including human and murine endometrium.

Asherman's Syndrome (AS) is characterized by intrauterine adhesions and is associated with infertility due to loss of normal endometrium. Hysteroscopy is the gold standard of methods for diagnosis of these intrauterine adhesions. However, it has certain potential complications such as uterine perforation and the possibility of adhesion recurrence in moderate and severe cases.

Therefore, stem cell therapy targeting the endometrium with the aim of replacing the damaged tissue, offers a promising approach for treating AS and Endometrial atrophy (EA). In a pilot trial, our research group demonstrated, for the first time, that CD133+ BMDSC autologous cell therapy may be useful in treating patients with AS and EA and a wish to conceive. These cells are capable of inducing proliferation of the neighbouring endometrial cells in the damaged endometrium. Given these results, the European Medicines Agency (EMA) approved the designation of orphan drug (ODD) to the investigational product IGX1 (treatment with autologous CD133+ stem cells) for the experimental treatment of Asherman's Syndrome (EMA/OD/313/16).

Based on these previous facts, a phase I/II clinical trial "ENTIRE" (code IGX1-ENT-XS-16-01 and European Union Drug Regulating Authorities Clinical Trials -EudraCT- number 2016-003975-23) was designed.

In order to study relevant effects of stem cell therapy in AS and respond to the clarifications requested by the AEMPs (Agencia Española de Medicamentos y Productos Sanitarios), the main objective of the present study is to evaluate the safety, tolerability, as well as the biodistribution, expression and cellular characterization of IGX1 (CD133+ cells selected after mobilization and collection of peripheral blood progenitor cells - CPSP) in a murine model with Asherman-induced Syndrome (preclinical study). In addition, other possible endothelial and blood markers of this cellular subpopulation will be characterized by flow cytometry, as well as the viability and potency of these cells.

ELIGIBILITY:
Inclusion criteria:

1. Donors of of hematopoietic stem cells whose written informed consent approved by the Ethics Committee (EC) has been obtained, after having been duly informed of the nature of the study and voluntarily accepted to participate after being fully aware of the potential risks, benefits and any discomfort involved.
2. Women of reproductive age between 18-44 years old (both inclusive).
3. BMI: 18-30 Kg/m2 (both inclusive)
4. Adequate hepatic and renal function defined as:

   * Total bilirubin <1.5x Higher Normal Validity (VSN)
   * Aspartate aminotransferase (AST) and Alanine aminotransferase (ALT) <2.5x VSN and
   * Serum creatinine <1.0 mg/dl; if the serum creatinine is >1.0 mg/dl, the estimated glomerular filtration rate (EGF) should be >60 ml/min/1.73 m2.
5. Absence of severe cardiac pathology.
6. Negative blood pregnancy test.
7. Eastern Cooperative Oncology Group (ECOG) = 0-1.
8. Negative serology for HIV, HCV, HBSAg, HBcAg and Syphilis (recent <30 days).
9. Normal coagulation study.
10. Adequate peripheral venous access.
11. Absence of serious psychiatric illness.
12. Ability of the donor to understand and comply with the study procedures.

Exclusion Criteria:

1. Absence of peripheral venous access.
2. Patients who have participated in another clinical trial or have received an investigational treatment during the last 30 days, unless the sponsor approves it.
3. Existence of serious or uncontrolled bacterial, fungal or viral infections that, could interfere with the participation of the donor in the study or in the evaluation of the results.
4. Any disease or unstable medical condition that may endanger the safety of the donor and their compliance with the study. (i.e., previous or current oncological or hematological diseases).

Ages: 30 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 5 (Estimated)
Dates: Start 2018-07-27 (Actual); Primary Completion 2019-10 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Number of CD133+ | 0 hours
  Total number of CD133+ obtained after the apheresis
Polymorphonuclear cells | 0 hours
  Total number of polymorphonuclear cells obtained

SECONDARY OUTCOMES:
Percentage of viable cells | 0 hours, 3 hours and 18 hours
  Evaluation of cell viability
Number of Colony-forming unit (CFU) | 0 hours, 3 hours and 18 hours
  The number of viable bacteria or fungal cells in the sample
Concentration of Pathogens | 0 hours
  Cells culture and gram stain
Expression of hematopoietic stem cells (subtypes: CD133+, CD56+, CD66+, CD14+, CD19+, CD3+, CD45+, CD34+) | 18 hours from extraction
  Isolation stem cells by Fluorescence Activated Cell Sorting Cytometry (FACS)

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Santamaria, MD PhD, Principal Investigator — Hospital Vall d'Hebron
Locations (1):
- Hospital Vall D´Hebron, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No